CLINICAL TRIAL: NCT04059835
Title: OptiBra Study, Optimal Postoperative Bra After Breastcancer Surgery - an RCT
Brief Title: OptiBra Study, Optimal Postoperative Bra After Breastcancer Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Backman, Medicine Doctor, Oncologynurse, Karolinska University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: KarolinskaUD
Record Dates: First submitted 2019-07-26; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Bra; Breast Cancer Surgery; Complication; Compression; Symptoms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial two Groups
Masking Description: Not blinded but randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard (Active Comparator): Standard bra, soft
  Interventions: Other: OptiBra study
- compression bra (Experimental): experimental bra, compression and stabile
  Interventions: Other: OptiBra study

INTERVENTIONS:
Other: OptiBra study — compare two different bra after breast cancer surgery

SUMMARY:
This study evaluates how two different types of postoperative bra 1) standard bra, soft VS 2) compression bra compression after breast cancer surgery affect pain, seroma, other symptoms and complications, and the womans experience of comfort

DETAILED DESCRIPTION:
Background

Breast cancer is the most common form of cancer in women and in Sweden about 9700 women are affected each year.Therefore, it is of great importance to promote the rehabilitation process by minimizing unnecessary symptoms and complications that may arise during a breast cancer treatment. Surgery is the primary cure for breast cancer and about 40% need to undergo a major surgical procedur and major operations also involve an increased risk of complications and symptoms.

Pain is the most common reported symptom in women who are operated on for breast cancer other complications after surgery that may occur are seroma, wound infektions and swelling.

No published evidence exists for the benefit and effect in pain relief from wearing a bra as a support after breast surgery is available, therefore it is important to evaluate useful and simple methods that the patient can manage herself that can minimize the experience of pain and other symptom after breast cancer surgery.

At Karolinska University Hospital's breast cancer center, women who undergo breast surgery are offered a bra after surgery in order to provide good support for the patient to feel safe, comfortable and minimize complications and symptoms such as pain. Two different types of bra are used and, according to the clinical staff at Karolinska's breast cancer center clinical experience, there is disagreement about which type of bra gives the optimal effect in different surgical procedures to reduce symptoms and post-operative complications. Neither is there enough knowledge about and how women experience comfort from the bra they received from the healthcare, which is important as the bra should be used large parts of the day for about 3 weeks after the procedure. Lack of knowledge makes it difficult to provide person-centered care for each individual. The purpose of this study is to compare two different types of bra after breast cancer surgery and to evaluate whether a particular type of bra affects the perception of pain, other symptoms, the occurrence of complications and experiences of bra comfort.

Purpose

To compare two different types of postoperative-bra after breast cancer surgery and to evaluate how a particular type of bra affects the perception of pain, other symptoms, the occurrence of complications and comfort.

Outcome Measure

The primary outcome measure is the presence of pain. Secondary outcome measures are, other symptoms, seroma, wound complications, and the patient's experience of satisfaction with support and comfort when using their postoperative bra.

Design

Randomized controlled trial aimed to comparing two groups of women undergoing breast cancer surgery.

Participant

Women diagnosed with breast cancer and undergoing breast surgery.

Data Collection

The data collection will take place at the Breast Center, Karolinska University Hospital in Solna, where approximately 500 breast cancer operations are performed every year. The women will be identified by the nurse or doctor at the MDT conference. The identified women will be asked about the participation of the nurse / doctor at the new visit to the surgeon's reception and bring written information home with them about the study. A few days after the new visit, the woman is called by a researcher or nurse for further oral information and the women who wish to participate will be given written informed consent. After this, baseline measurement and randomization are performed to one of two groups. Evaluation will be performed on two occasions, prior to surgery (baseline for pain and other symptoms, demographic issues) and 3 weeks after surgery (pain, symptoms, clinical assessment of the breast). Demographic (age, education, etc.) and medical information (weight, BMI, illness history, smoking, alcohol habits and physical activity, etc.) as well as the type of surgical procedure and drain are collected through medical records.

Inclusion

Women from 18 years of age with malignant tumor of the breast gland to undergo surgery.

Exclusion

Men with breast cancer. Women with benign tumors or women with health factors where the assessment is that Bra use from healthcare is not necessary or possible.

Compliance and instruments

The participant will be instructed to use the bra according to. Instruction and adherence to intervention will be via diary pages where the participant for 3 weeks briefly fills in (number of days) and how often (number of hours / day) you have used the bra you received from the health care. Primary outcome measure is; pain, secondary outcome measures are, presence of seroma, symptoms after breast surgery mainly swelling, redness, and satisfaction with the use of bra focusing on comfort and support. Instruments for self-estimated outcome measures that will be used are;

* To measure the perception of pain comes the estimation instrument VAS (visual analogue scale). VAS is a 10 cm long horizontal line where on one side measures "no pain" and on the other "worst possible pain" and the patient places a mark on the line corresponding to the perceived pain .
* To measure chest symptoms, EORCT QLQ-BR 23 will be used. BR 23 is a questionnaire that measures common symptoms of breast cancer disease and treatment (eg you have had difficulty lifting or moving your arm, have you had pain around your breast).
* The presence of wound complications, seroma and other symptoms reported by the patient (swelling, redness) will be assessed by clinical assessment of the nurse and medical record. E.g. Seroma will be assessed on the basis of a template based on the number of drops and the amount / ml of dropped liquid.

To examine how participants experience the convenience, comfort, and support of the postoperative bra they used in the study, participants will answer study-specific questions (open and closed) regarding patient experience (patient satisfaction) regarding BRA use that relates to comfort, support and comfort.

Intervention

Participants are randomized into one of two groups. Group 1) is offered the more stable bra with some compression after breast cancer surgery, while Group 2) is offered a softer bra without compression. Participants are encouraged to use the bra according to instructions and record the number of hours / days for use in a diary. When returning to a nurse / doctor after about 3 weeks of use, all participants respond to survey questions about pain, other symptoms and experience of support and comfort during use, and undergo a clinical assessment of the nurse according to a template with respect to seroma, number of taps, quantity and occurrence of complications (eg wound infection). Compliance with intervention takes place trough a simple diary which participants fill in for 3 weeks eg. how long (number of days) and often (number of hours / day) have you used the bra you received from the healthcare system, as well as grading daily pain according to the VAS- scale.

To determine if there are differences between 2 groups with respect to the variable pain as the primary outcome measure, a sample size of 80 women per group is calculated to be necessary with a power of 0.80 percent and a significance level of <0.05. Given that subgroup analyzes (about 5 groups - mastectomy +- SN, mastectomy +- axillary, sector + - SN, sector +- axillary and primary reconstruction) will be done and a planned 10% drop-out, 100 women per group will be included.

Analysis

Quantitative data will be processed using relevant statistical parametric methods for normally distributed data and non-parametric methods for non-normally distributed data. Analyzes will investigate differences between groups as well as within the group (ANOVA) as well as analyzes for the relationship between different parameters (eg type of bra and surgical procedure). Demographic baseline data is reported as descriptive statistics (SD, mean, frequency). Statistics will be used for support.

Ethical issues

The current research project will follow the basic ethical principles that include the information requirement, the consent requirement, the confidentiality requirement and the use requirement . Involved persons in the team for the BH study all have long experience of meeting people with cancer diagnosis. Close ethical discussion with expertise in the research group on the routines that exist today for bra use after surgery and in randomization so as not to cause or risk injury to the woman. All participants will; receive oral and written information about the study, have the opportunity to ask questions via telephone or mail during the entire study period (the information requirement). Participants will be informed that participation is completely voluntary and that there is no disadvantage if participation is canceled (the consent requirement). Personal data will be de-identified and handled in accordance with statutes to minimize the identity of the participants for unauthorized persons in the reporting of results (the confidentiality requirement).

The collected data will only be used for research purposes (the use requirement).

ELIGIBILITY:
Inclusion Criteria:

Women from 18 years

Malignant tumor of the breast gland to undergo surgery.

Exclusion Criteria:

Men with breast cancer Women with benign tumors Women with health factors where the assessment is that BRA use is not necessary or possible.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measure | 21 days from operations day
  VAS scale ( Visual analoge scale) , each item is score, 0= no pain to 10= pain as bad as can be. yielding at total between 0 and 10

SECONDARY OUTCOMES:
Postoperative breastsymptoms | report every day, 21 days after operation
  Clinical observation by doktor 3 weeks after surgery and Medical records
Seroma | This will be examine 21 days after the surgery at the revisit to surgon
  Clinical observation by doktor registrated in Medical journal about number of dropping and ml each dropping. And % of patients suffering from seroma after surgery
Patients experience of symptoms and comfort | Reported basline and 21 days after operation
  EORTC QLQ BR23 questionnaire measure symptoms after breascancer surgery, a 4 item scale, each item i scored from -not at all to verry mutch. We will follow the EORTC QLQ manual for calculation, scale 1-100, where high scores mean more severe symptoms And some study specific questions about experience of Comfort ex.have you experienced that the BRA has given you support
Pain medication intake after surgery | Report every day, 21 days after operation
  Self care-diary

CONTACTS AND LOCATIONS:
Overall Officials: Malin Backman, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fallbjörk U, Salander P & Rasmussen BH. From
- [Derived] Backman M, Hassan-Nur M, Fridblom K, Johansson H, Fredholm H, Fredriksson I. OptiBra study, a randomized controlled trial on optimal postoperative bra support after breast cancer surgery. Eur J Oncol Nurs. 2023 Apr;63:102285. doi: 10.1016/j.ejon.2023.102285. Epub 2023 Feb 15. PMID 36893575